CLINICAL TRIAL: NCT02774213
Title: An Observational Study to Collect Data Characterizing Analgesia in Patients Suffering From Bone Metastasis Induced Pain
Brief Title: A Study to Collect Data About Analgesia in Patients With Bone Metastasis
Status: Completed | Type: Observational
Sponsor: Tools4Patient (Other)
Responsible Party: Sponsor
Other Study IDs: T2001-01
Record Dates: First submitted 2016-04-20; First posted 2016-05-17 (Estimated); Results first posted 2019-08-19 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-07

CONDITIONS: Bone Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Use of potentially available archived tumor tissue block and/or aliquot of standard safety laboratory blood sample for genotyping purposes are optional in this study for patients recruited in Belgium.
  This optional research is not proposed to any patient recruited in France
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Questionnaires completion
Other: Clinical Pain Assessments

SUMMARY:
Up to 180 patients with bone metastasis and requiring analgesic treatment will be followed during 4 to 10 weeks. All patients will continue to receive their cancer therapeutic treatments and be treated for pain relief exactly as they would normally be by the Investigator based on their needs. During their regular visits to the Investigator, patients will complete questionnaires and Clinical Pain Assessments.

ELIGIBILITY:
Inclusion Criteria:

* Patients with bone tumors or bone metastasis from any primary cancer origin that is supported by histological or radiological investigations.
* Patients having been or being treated for their bone metastasis and/or their primary cancer.
* Patients who require analgesic treatment for unsatisfactory pain relief.
* Patients will be required to score at least 4 on the WAPS 11-point NRS during the week preceding enrollment.
* Patients undergoing or not a radiotherapy program provided visit procedures are performed before any radiotherapy sessions if scheduled on the same visit days.
* Are men or women of at least 18 years of age.
* Are reliable and willing to make themselves available for the entire duration of the study and are willing to follow study procedures.
* Have given written informed consent approved by the relevant Ethics Committee governing the study site.

Exclusion Criteria:

* Patients having had a major surgery within 28 days prior to signing Informed Consent Document or planning to have a major surgery during the study.
* Patients having a life expectancy < 3 months according to Investigator judgment.
* Patients having poor nutritional status or whose condition is unstable or who could be rapidly deteriorating in such a way that they would not be able to complete the study.
* Patients with a current or recent history unrelated to their cancer condition, as determined by the Investigator, of severe, progressive, and/or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurological, or cerebral disease which would interfere with the patient's participation in the study.
* Patients having a Karnofsky performance status below 70% or WHO score (Eastern Cooperative Oncology Group (ECOG)/Zubrod score) above 1.
* Are Investigator site staffs directly affiliated with this study and/or their immediate families. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
* Any other relevant medical disorder likely to interfere with the trial or represent a risk for the patient.
* Patients under legal protection, according to the country law.
* Patients currently enrolled in a clinical trial involving use of an investigational drug or device, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study, or in an exclusion period according to the national law.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 180 patients diagnosed with bone metastasis suffering from pain will be enrolled into the study to have up to approximately 140 completers
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2014-07; Primary Completion 2017-04-28 (Actual); Study Completion 2017-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro Pereira, Study Director — Tools4Patient
Locations (8):
- Belgium (4):
  - Institut Bordet, Brussels
  - Cliniques Universitaires Saint Luc, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - ATC, CHU Sart Tilman, Liège
- France (4):
  - Hôpital A. Mignot, Le Chesnay
  - Centre Oscar Lambert, Lille
  - Hôpital La Timone, Marseille
  - Institut Curie, Paris

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cancer-Induced Bone Pain (CIBP): Cancer patients with bone metastasis suffering from pain
Period: Overall Study
Arm/Group | Cancer-Induced Bone Pain (CIBP)
Started | 74
Completed | 55
Not Completed | 19

BASELINE CHARACTERISTICS:
Arm/Group | Cancer-Induced Bone Pain (CIBP)
Number analyzed (Participants) | 74
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 60.1 [54 to 67]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Only subjects completing the study per protocol were analysed
  Participants
    number analyzed (Participants) | 53
    Female | 42
    Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Patient's Change From Baseline of Pain Severity, as Measured by the Weekly Means of the Daily Average Pain Scores (APS)
Description: 11-point Numeric Rating Scale from 0 to 10 with 0 meaning no pain and 10 pain as bad as you can imagine; baseline measure was the Weekly Average Pain Score (WAPS), over the week first visit (the last 7 days); end of study measure was the mean of the APS of the last 7 days prior to last visit (Visit 2)
Time Frame: Time zero equals baseline up to after at least 4 weeks of observation (Visit 2)
Population: Only the patients completing the study per protocol were analyzed. APS was available for 47 patients amongst the per protocol completers.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cancer-Induced Bone Pain (CIBP)
Number analyzed (Participants) | 47
units on a scale | 2.26 (2.95)

2. Secondary Outcome: Patient's Change From Baseline of Pain Severity, as Measured by the Weekly Means of the Daily Worst Pain Score (WPS)
Description: 11-point Numeric Rating Scale from 0 to 10 with 0 meaning no pain and 10 pain as bad as you can imagine; baseline measure was was the mean of the WPS of the first 7 days after first visit (Visit 1); end of study measure was the mean of the WPS of the last 7 days prior to last visit (Visit 2)
Time Frame: Time zero equals baseline up to after at least 4 weeks of treatment (Visit 2)
Population: Only the patients completing the study per protocol were analyzed. WPS was available for 46 patients amongst the per protocol completers.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cancer-Induced Bone Pain (CIBP)
Number analyzed (Participants) | 46
units on a scale | 1.23 (2.07)

3. Secondary Outcome: Patient's Change From Baseline of Pain Severity as Measured by the Brief Pain Inventory (BPI)
Description: The pain severity score of BPI is an arithmetic average of the 4 severity scores reported on an 11- point NRS going from 0 (no pain) to 10 (pain as bad as you can imagine).
  The BPI severity questions are:
  3. Your pain at its worst in the last 24 hours? 4. Your pain at its least in the last 24 hours? 5. Your pain on the average? 6. How much pain you have right now?
Time Frame: Time zero equals baseline up to after at least 4 weeks of treatment (Visit 2)
Population: Only the patients completing the study per protocol were analyzed. APS was available for 51 patients amongst the per protocol completers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cancer-Induced Bone Pain (CIBP)
Number analyzed (Participants) | 51
score on a scale | 1.16 (2.11)

4. Secondary Outcome: Patient's Change From Baseline of Investigator Global Assessment of Changes (IGAC)
Description: Investigator subjective evaluation of patient condition using an 11-point NRS with 0 meaning best and 10 worst
Time Frame: Time zero equals baseline up to after at least 4 weeks of treatment (Visit 2)
Population: Only the patients completing the study per protocol were analyzed. IGAC was available for 48 patients amongst the per protocol completers.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cancer-Induced Bone Pain (CIBP)
Number analyzed (Participants) | 48
units on a scale | 1.31 (2.42)

5. Secondary Outcome: Patient's Change From Baseline of Patient Global Assessment of Changes (PGAC)
Description: Patient subjective evaluation of patient condition using an 11-point NRS with 0 meaning best and 10 worst
Time Frame: Time zero equals baseline up to after at least 4 weeks of treatment (Visit 2)
Population: Only the patients completing the study per protocol were analyzed. PGAC was available for 50 patients amongst the per protocol completers.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cancer-Induced Bone Pain (CIBP)
Number analyzed (Participants) | 50
units on a scale | 1.22 (2.64)

6. Secondary Outcome: Patient's Change From Baseline of Pain Intensity Measured After Clinical Pain Assessments (CPAs)
Description: Number of symptoms measured after Clinical Pain Assessments (CPAs), 0 no symptom to 3 all the three symptoms : Hyperalgesia, Hypoesthesia, and Sensory loss.
Time Frame: Time zero equals baseline up to after at least 4 weeks of treatment (Visit 2)
Measure: Mean (Standard Deviation); unit: Number of symptoms
Arm/Group | Cancer-Induced Bone Pain (CIBP)
Number analyzed (Participants) | 67
Number of symptoms | 0.34 (0.57)

7. Secondary Outcome: Patient's Change From Baseline of Quality-of-Life Questionnaire in 30 Questions (QLQ-C30).
Description: Pain scale of the Quality-of-Life Questionnaire in 30 questions (QLQ-C30); 2 items in the Pain scale ranging each from 1 to 4 (high score for a symptom scale / item represents a high level of symptomatology / problems); Pain score is sum of of the 2 items
Time Frame: Time zero equals baseline up to after at least 4 weeks of treatment (Visit 2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cancer-Induced Bone Pain (CIBP)
Number analyzed (Participants) | 51
score on a scale | -5.99 (13.81)

8. Secondary Outcome: Patient's Change From Baseline of Pain Interference as Measured by the Brief Pain Inventory (BPI)
Description: The pain interference score of BPI is an arithmetic average of the 7 interference scores reported on an 11-point NRS going from 0 (does not interfere) to 10 (completely interferes)
  The BPI interference questions are:
  9. Pain has interfered in the last 24 hours with
  1. General Activity?
  2. Mood?
  3. Walking Abililty?
  4. Work?
  5. Relations with other people?
  6. Sleep?
  7. Enjoyment of life?
Time Frame: Time zero equals baseline up to after at least 4 weeks of treatment (Visit 2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cancer-Induced Bone Pain (CIBP)
Number analyzed (Participants) | 51
score on a scale | 1.42 (2.55)

ADVERSE EVENTS:
Time Frame: Not applicable: observational study (no safety measurements)
Description: Not applicable: observational study (no safety measurements)
Arm/Group | Cancer-Induced Bone Pain (CIBP)
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-04-10): https://cdn.clinicaltrials.gov/large-docs/13/NCT02774213/SAP_000.pdf
  • Study Protocol (2014-11-24): https://cdn.clinicaltrials.gov/large-docs/13/NCT02774213/Prot_001.pdf